CLINICAL TRIAL: NCT01921504
Title: Effect of Acupuncture on Patients With Functional Dyspepsia: a Multi-center, Randomized, Waitlist-controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Acupuncture and Meridian Science Research Center (Other)
Responsible Party: Principal Investigator, Jae-Woo Park, Associate Professor, Department of Korean Internal Medicine, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHNMC-OH-IRB 2013-006
Record Dates: First submitted 2013-08-07; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Acupuncture; Genotype; Ghrelin
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Participants in this group are given twice-a-week acupuncture treatment for 4 weeks.
  Interventions: Device: Acupuncture
- No treatment (No Intervention): The participants in this group are supposed to wait without any intervention for first 4 weeks. Then they receive the identical acupuncture treatments as in the treatment group for the following 4 weeks.

INTERVENTIONS:
Device: Acupuncture — Acupuncture treatment
  1. Acupuncture rationale 1a) Style of acupuncture: body acupuncture (in accordance with meridian theory)
  2. Needling details 2a) Number of needle insertions per subject per session: 9-19 2b) Acupoints: Basic points - Large Intestine(LI)4, Stomach(ST)36, Liver(LR)3, Spleen(SP)4, Conception Vessel(CV)12 Optional points - Gallbladder(GB)21, Small Intestine(SI)14, Pericardium(PC)6, External points of Hand and Neck(EX-HN)5, Stomach(ST)34 2c) Depth: 5 ~ 30mm 2d) Response sought: 'Deqi' 2e) Needle stimulation: Manipulation 2f) Retention time: 15 minutes 2g) Needle type: 25 X 30 mm, sterilized stainless steel needle, Dongbang Inc., Korea
  Other Names: Acupuncture treatment
  Arms: Acupuncture

SUMMARY:
The aim of the study is to investigate the effect of acupuncture treatment on functional dyspepsia.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a functional gastrointestinal disorder without any structural lesion. FD is claimed to affect 25% of the population in South Korea. Although conventional approaches based on current evidence such as proton pump inhibitor and prokinetic agents have been used, many FD patients turn to traditional Korean Medicine treatment largely due to the lack of satisfactory effect of these treatments.

Acupuncture treatment, one of the most sought therapeutic modalities in traditional Korean Medicine, has been commonly used for gastrointestinal disorders in Korea. However, the effect of acupuncture on FD has not been rigorously evaluated. In the present study, we will investigate whether 8 sessions of acupuncture treatment over 4 weeks, in comparison with no acupuncture treatment, i.e. waitlist-control, improve symptoms of FD. Outcome measures include proportion of responder, Korean version of Nepean Dyspepsia Index, EuroQol-5 Dimension, Functional Dyspepsia-Related Quality of Life, Beck's Depression Inventory, State-Trait Anxiety Inventory and ghrelin hormone. Genome-wide association study (GWAS) will be also conducted to elucidate any possible difference in genotype between responders and non-responders to acupuncture treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 ~ 75, with a elementary-school diploma or higher, should be able to read and write Korean
* One who meet Rome III FD criteria* and has been suffering from FD for the last 3 months with symptom onset at least 6 months prior to diagnosis

  * One or more of the following:

    1. Bothersome postprandial fullness
    2. Early satiation
    3. Epigastric pain
    4. Epigastric burning
* One who checks more than 4 points on visual analogue scale (VAS) for dyspeptic symptoms
* One who has normal esophagogastroduodenoscopy results within a year and been diagnosed with FD by a specialist consultation
* One who receives no other treatments during the study
* One who voluntarily agrees with study protocol and signs an written informed consent

Exclusion Criteria:

* One who has peptic ulcer or gastroesophageal reflux disease (GERD)
* One who has obvious signs of irritable bowel syndrome (IBS)
* One who has alarm symptoms (weight loss, black or tar stool, dysphagia)
* One who has serious structural disease (disease of heart, lung, liver or kidney) or mental illness
* One who has had surgery related with the gastrointestinal tract (Appendectomy more than 6 months ago is acceptable)
* One who is pregnant or breastfeeding
* One who is taking drugs which might affect gastrointestinal tract (Wash-out period: 2 weeks before participating in the trial)
* One who is HIV-positive
* One who has a problem of malabsorption or maldigestion
* One who has difficulties in attending the trial or receiving treatments (e.g Paralysis, serious mental illness, dementia, drug addiction, busyness, severe disorder in vision or hearing, impossibility of visit, illiterate, etc.)
* One who does not want to sign the informed consents
* One who has clotting disorders or leukopenia, pace-maker, seizure disorders or is taking anticoagulant therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders | Once in treatment period (4 wks)
  The proportion of patients who answer "Yes" to more than half of adequate relief questions in the treatment period.
  Patients are expected to report their response to the acupuncture treatment by answering the following question at each visit: "After the last visit, have you had adequate relief of your stomach pain or discomfort?" Questions will be asked at each visit during treatment period (Twice a week for 4 wks, total 8 times - 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4 wks). Responders are defined as patients reporting adequate relief for at least 50% of the study period (more than 4 times of "Yes" to adequate relief question out of total 8 questions). The proportion of responder will be compared statistically between experimental group and no intervention group.

SECONDARY OUTCOMES:
Nepean Dyspepsia Index - Korean version (NDI-K) | After treatment (4 wks)
  The Nepean Dyspepsia Index is a reliable and valid measure of quality of life in FD. The Nepean Dyspepsia Index originally contains 42 items designed to measure impairment of a subject's ability to engage in relevant aspects of their life because of dyspepsia. It was subsequently shortened to 25 items, yielding 5 sub-scales. NDI-K, validated in 2004 by Choi at al., made up of 2 sections which are about symptom-based questions and quality of life. In this trial, symptom-based questions, i.e. questions about period, severity and distressful degree of 15 symptoms, will be evaluated.
EuroQol-5 Dimension (EQ-5D) | After treatment (4 wks)
  EQ-5D is a standardized instrument as a measure of health outcome. EQ-5D consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  First page is made up of 5 questions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each question has 3 levels: no problem, some problems, major problems.
  Second page consists of EQ VAS and its explanation. EQ VAS records the respondent's self-rated health on a vertical visual analogue scale where each endpoint is labelled either 'Best imaginable health state' and 'Worst imaginable health state'.
Functional Dyspepsia-Related Quality of Life (FD-QoL) Questionnaire | After treatment (4 wks)
  The FD-QOL scale is a 21-item Likert-type questionnaire that can easily be completed within 5 min. Short administration time and high comprehensibility supports the feasibility of measuring health-related quality of life.
Beck's Depression Inventory (BDI) | After treatment (4 wks)
  The Beck Depression Inventory (BDI), created by Dr. Aaron T. Beck, is a 21-question multiple-choice self-report inventory and one of the most widely used instruments for measuring the severity of depression.
The State-Trait Anxiety Inventory (STAI) | After treatment (4 wks)
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety (anxiety triggered by a specific event), and trait anxiety (anxiety derived from personal characteristic). Higher scores are positively correlated with higher levels of anxiety.
Ghrelin hormone measurement (1. Total ghrelin, 2. Deacylated ghrelin) | After treatment (4 wks)
  Ghrelin is a gut-derived peptide found in the stomach. It is known to play a role in the regulation of gastric motility and appetite.
Genotype analysis by Axiom® exome genotyping arrays | First visit (0 wk)
  Genome-wide association study (GWAS)examines genetic variants in different individuals to see if any variant is associated with a trait. In this study, the GWAS is planned to elucidate any associations between genetic difference and response to acupuncture treatment in FD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-woo Park, Doctor's degree, Principal Investigator — Kyung Hee University Hospital at Gangdong, Seoul, Repulic of Korea
Locations (2):
- South Korea (2):
  - Kyung Hee University Oriental Medicine Hospital, Seoul, Dongdaemun-gu
  - Kyung Hee University Hospital at Gangdong, Seoul, Gangdong-gu

REFERENCES:
- [Derived] Han G, Ko SJ, Park JW, Kim J, Yeo I, Lee H, Kim SY, Lee H. Acupuncture for functional dyspepsia: study protocol for a two-center, randomized controlled trial. Trials. 2014 Mar 22;15:89. doi: 10.1186/1745-6215-15-89. PMID 24655542
- See also: Acupuncture and Meridian Science Research Center (AMSRC) — http://amsrc.khu.ac.kr/center/center_03_eng.php